CLINICAL TRIAL: NCT01034215
Title: Multi-Media Imagery Program for Breast Cancer Patients (Phase II)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mind Matters Research LLC (Other)
Responsible Party: Lynda Freeman, Ph.D., Principal Investigator and CEO, Mind Matters Research LLC, Mind Matters Research LLC
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: MMR-117597
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2009-12

CONDITIONS: Breast Cancer
Keywords: Behavioral; Quality of Life; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Imagery Practice, live trainer (Active Comparator): Patients attend a five week training program, with the instructor in the room with them, and actively practice imagery techniques, both in the classroom, and daily, outside of the classroom. Classes are four hours a week for five weeks. Patients practice what they learn for a full 17 weeks, beginning with the first week of class.
  Interventions: Behavioral: Envision the Rhythms of Life Program
- "Envision the Rhythms of Life" /video (Active Comparator): Patients learn to practice passive, active and targeted imagery for the purpose of improving mood state, modifying physiology (HRV, Body temperature, pain reduction) and also to mitigate the effects of their treatments, as defined by the IOM: chemo brain, fatigue, sleep deprivation, stress, anxiety, depression, and/or PTSD.
  Interventions: Behavioral: Envision the Rhythms of Life Program/Distance
- Waitlist Control Group (No Intervention): No treatment delivery during the 17 weeks of testing live delivery (trainer in the room with patients) vs. distance delivery (trainer delivers program via telemedicine/videoconferencing equipment)

INTERVENTIONS:
Behavioral: Envision the Rhythms of Life Program — Patients learn to practice passive, active and targeted imagery for the purpose of improving mood state, modifying physiology (HRV, Body temperature, pain reduction) and also to mitigate the effects of their treatments, as defined by the IOM: chemo brain, fatigue, sleep deprivation, stress, anxiety, depression, and/or PTSD. Program is delivered with trainer present in the room.
  Other Names: Envision the Rhythms of Life, Live delivery
  Arms: Imagery Practice, live trainer
Behavioral: Envision the Rhythms of Life Program/Distance — Patients learn to practice passive, active and targeted imagery for the purpose of improving mood state, modifying physiology (HRV, Body temperature, pain reduction) and also to mitigate the effects of their treatments, as defined by the IOM: chemo brain, fatigue, sleep deprivation, stress, anxiety, depression, and/or PTSD. Program is delivered by videoconference equipment
  Other Names: Envision the Rhythms of Life Program, Distance Delivery
  Arms: "Envision the Rhythms of Life" /video

SUMMARY:
Global Objective: To improve quality of life and reduce stress for breast cancer survivors. To address the late-term and long-term effects of breast cancer treatment, as defined by the Institute of Medicine, including chemo brain, fatigue, sleep deprivation, stress, anxiety, depression, and PTSD.

Phase II Aims: (1) To demonstrate the clinical efficacy (i.e., improved quality of life, stress reduction, participant satisfaction with product) of the "Envision the Rhythms of Life" program and (2) to establish the technical merits of the program's distance-delivery (videoconferencing hardware and software) and instructional technology (i.e., animations, graphically enhanced PowerPoint instructional materials, full-color program manuals, art-as-imagery, and audio-imagery). "Envision the Rhythms of Life" instructs breast cancer survivors in the practice of individualized, emotionally supportive, and biologically accurate imagery and consists of 5, 4-hour long, interactive classes and between-class instructor support.

Instructional Options: Option 1 delivers the program technology (animations, PowerPoint, manuals, art, audio-art) with instructor and participants in the same room. Option 2 delivers the program at-a-distance, to a small group of, via videoconferencing software and camera systems (Alaska and Seattle) to low, moderate or high bandwidth areas. Each option delivers program three times (total of 45 participants for each option). A website portal provides all program information and materials.

Design and Method: Program will be delivered to 135 breast cancer survivors who have completed conventional care (surgery, radiation, IV chemotherapy) for at least six weeks. Differences in option 1 and 2 outcomes will be compared to each other and to controls; combined outcomes of option 1 and 2 will be compared to controls; and waitlist control outcomes will be compared to their extended baseline. Hypothesis: Options 1 and 2 will both produce significantly better outcomes than waitlist control group.

DETAILED DESCRIPTION:
DESCRIPTION: To improve quality of life and reduce stress for breast cancer survivors. Phase II Aims: (1) To demonstrate the clinical efficacy (i.e., improved quality of life, stress reduction, participant satisfaction with product) of the "Envision the Rhythms of Life" program and (2) to establish the technical merits of the program's distance-delivery (videoconferencing hardware and software) and instructional technology (i.e., animations, graphically enhanced PowerPoint instructional materials, full-color program manuals, art-as-imagery, and audio-imagery). "Envision the Rhythms of Life" instructs breast cancer survivors in the practice of individualized, emotionally supportive, and biologically accurate imagery and consists of 5, 3-hour long, interactive classes and between-class instructor support. Instructional Options: Option 1 delivers the program technology (animations, PowerPoint, manuals, art, audio-art) with instructor and 15 participants in the same room. Option 2 delivers the program at-a-distance, to a small group of 15, via videoconferencing software and camera systems (Alaska and Seattle) to low, moderate or high bandwidth areas. Each option delivers program three times (total of 45 participants for each option). A website portal provides all program information and materials. Design and Method: Program will be delivered to 135 breast cancer survivors who have completed conventional care (surgery, radiation, IV chemotherapy) for at least six weeks. Differences in option 1 and 2 outcomes will be compared to each other and to controls; combined outcomes of option 1 and 2 will be compared to controls; and waitlist control outcomes will be compared to their extended baseline. Long-Term Objectives: This innovative project integrates technology with bandwidth-sensitive multi-media conferencing strategies to deliver a virtual mind-body, imagery intervention. The technology will allow seamless program delivery to interested survivors across the country during Phase III. Instructional technology, designed per Phase I participant feedback, will serve to 'jump-start' potent imagery practice and will optimize clinical efficacy. Commercial application and survivor participation is not limited by location, work schedule, or health status, addressing issues of barriers to access of care. Although desirable, instructional options 1 and 2 do not require survivors to have computer skills or internet access. The program is designed to be culturally sensitive and supports individual spiritual practices. PUBLIC HEALTH RELEVANCE: This program addresses NCI and IOM summary reports that call for individualized supportive care for cancer survivors suffering disease-related distress. Changes in two disease-education program modules would allow the program to be used as supportive therapy for other forms of cancer across the country.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be a community-dwelling member 18 years of age or older. - The participant must be at least 18 because the assessment tools are not validated for use in minors.
* Participants should be able to read, write, and speak English.
* Participants must have been diagnosed with breast cancer and have completed surgery, which did not include Level III dissection of the axilla.
* Participants must obtain verification of diagnosis and treatment from their physician.
* Participants must agree to complete assessment instruments and take part in psychophysiological data gathering at baseline, 8 and 17 weeks and to provide required demographic information.
* Participants must sign informed consent, stating he/she understands the nature of the research and that he/she wishes to participate in the study. -
* Participants must agree to complete the required diaries, graphs and notebooks related to behavior assessment.
* Participants must display the ability to understand and respond to the assessment process and must demonstrate they are oriented to person, place, and time.
* Participants must agree to fully participate in all five imagery classes and to practice imagery skills for 20 minutes a day for 17 weeks.
* Participants must have completed major cancer treatment (i.e., surgery, and/or radiation and/or IV chemotherapy) for six weeks; participant must be visual and hearing capable.
* Oral chemotherapy does not preclude participation.

Exclusion Criteria:

* Participant will be excluded if he/she has a history of uncontrolled epileptic seizures.
* The investigators will exclude patients who cannot speak, read and write English.
* Patients will be excluded if they are not oriented to place, person, and time.
* Participants will be excluded if they have a major psychiatric diagnosis (schizophrenia, bi-polar disorder).
* The investigators will exclude patients who received a Level III dissection of the axilla.
* Participants will be excluded if they are visually or hearing impaired.
* Although imagery can be modified for the visually or hearing impaired, that model is significantly different from an imagery program for the visual and hearing capable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2008-08; Primary Completion 2010-09 (Actual); Study Completion 2011-10-11 (Actual)

PRIMARY OUTCOMES:
Primary Objective: Measure QOL differences between treatment groups: (delivered live vs videoconferencing) and as compared to the control group and their extended baseline. | Data is gathered at baseline (before intervention) and 8 weeks, and at 17 weeks.

SECONDARY OUTCOMES:
The secondary objective is for the purposes of improving program materials, documenting patient satisfaction, and recording patient experience of imagery. Focus groups, summary reports, and 10-point likert scales, rated from very dissatisfied (1) to very | Data gathered across each week, beginning with first week of intervention, for a period of 17 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lynda W Freeman, Ph.D., Principal Investigator — Mind Matters Research LLC
Locations (1):
- Gilda's Club Seattle, Seattle, Washington, United States

REFERENCES:
- See also: Website for "Envision the Rhythms of Life" cllinical trial and program — http://www.mindmattersresearch.com